CLINICAL TRIAL: NCT06542991
Title: An Open-label Study on the Clinical Efficacy of rTMS Intervention in PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Head, Dept of Neurology & Medical Psychology, Director, Cognitive Neuropsychology Lab, PRC, Anhui Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD-OPEN
Record Dates: First submitted 2024-08-03; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Transcranial Magnetic Stimulation; Parkinson Disease; Supplementary Motor Area
Keywords: Transcranial Magnetic Stimulation; Parkinson Disease; Supplementary motor area
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rTMS group (Experimental): On the basis of drug treatment, a course of TBS treatment is performed for 7 days.
  Interventions: Other: transcranial magnetic stimulation

INTERVENTIONS:
Other: transcranial magnetic stimulation — During treatment, the patient underwent cTBS targeting the left SMA for 7 consecutive days. Each treatment day comprised six rounds of cTBS, with a 15-minute interval between each. A single cTBS session involved trains of three pulses at 50 Hz, repeated every 200 ms (5 Hz), until reaching a total of 600 pulses, lasting 40s. Stimulation intensity remained at 80% of resting motor threshold. In total, patients received 25,200 pulses throughout the treatment period.

SUMMARY:
To demonstrate that intervention targeting the supplementary motor area (SMA) using precise navigation positioning can effectively improve motor symptoms in patients with Parkinson's disease.

DETAILED DESCRIPTION:
As an innovative non-invasive neuromodulation technology, repetitive transcranial magnetic stimulation (rTMS) has demonstrated efficacy in improving motor symptoms in patients with Parkinson's disease (PD). The supplementary motor area (SMA) has been identified as a brain region significantly associated with motor symptoms in PD patients. However, no large-sample clinical studies have yet established the clinical efficacy of rTMS, guided by neuroimaging navigation, targeting the SMA in patients with Parkinson's disease.

We describe a open-lable study designed to recruit 20 patients with idiopathic Parkinson's disease. Participants will be randomly assigned to receive either real stimulation or sham stimulation, with the left SMA undergoing 7 days of continuous theta burst stimulation (cTBS). The primary outcome measure is the change in the Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III scores from baseline to post-treatment and follow-up. Secondary outcomes include changes in scores on other clinical symptom scales.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥40 years old
2. Meet Movement Disorder Society standards;
3. Have no history of drug adjustment within 4 weeks before and during treatment;
4. The MDS-UPDRS Ⅲ score ≥8, and the Hoehn-Yahr rating is 1-4
5. MMSE ≥24，able to cooperate with the completion of behavioral tests and transcranial magnetic stimulation therapy.

Exclusion Criteria:

1. Head MRI/CT ruled out focal brain injury or severe leukoencephalopathy (Fazekas grade 3);
2. Various secondary parkinsonism syndromes (vascular parkinsonism, Parkinsonism combined with parkinsonism, drug parkinsonism, etc.);
3. Severe craniocerebral trauma, received craniocerebral surgery or deep brain stimulation treatment;
4. There are ferromagnetic implants in the body, such as cochlear implants, cardiac pacemakers, etc.
5. The person or first-degree relatives have a history of epilepsy, unexplained loss of consciousness, or are taking anticonvulsant drugs to treat epileptic seizures;
6. Diagnosed with a neuropsychiatric disorder other than PD
7. Have a history of drug abuse or drug use;
8. Participants in any clinical trial within the previous 6 month;
9. Pregnant/lactating women or subjects (including men) who have a birth plan within 6 months;
10. Other conditions deemed unsuitable for inclusion by the investigator.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale Part Ⅲ | baseline; day 8; week 5;week 9;
  The primary outcome was the change in MDS-UPDRS III from baseline to 9 weeks of follow-up. MDS-UPDRS III is a questionnaire used by uniformly trained professionals to evaluate motor symptoms in patients with Parkinson's disease[21]. The questionnaire consists of 18 items, which professionals need to score according to the patient's motor symptoms, on a scale of 0-4. Among them, items 3.3-3.8 and 3.15-3.17 can be divided into several sub-items according to the body parts. The results of MDS-UPDRS III are the total of 18 items.

SECONDARY OUTCOMES:
Hoehn-Yahr(H-Y) stage | baseline; day 8; week 5;week 9;
  It ranges from 1 to 5, and is evaluated based on the range of symptoms involved and whether balance is impaired in PD patients. The higher the score, the more severe the severity.
The timed up and go test | baseline; day 8; week 5;week 9;
  TUG measures in seconds how long it takes the subject to rise from the chair, walk 3 meters, turn around, walk back to the chair, and sit down. The test is often used to assess walking and balance in older adults. This also applies to evaluating the severity of walking and balance symptoms in patients with Parkinson's disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Cognitive Neuropsychology Lab Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No